CLINICAL TRIAL: NCT03473041
Title: Surgeon Tailored Hybrid Autologus Rectus Sheath Fascia Versus Midurethral Transobturator Tension Free Vaginal Tape For Treatment Of Stress Urinary Incontinence
Brief Title: Autologous Rectus Sheath Fascia Versus Midurethral Transobturator Tension Free Vaginal
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: sarah mohamed hassan (Other)
Responsible Party: Sponsor-Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 783
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Stress Urinary Incontinence
Keywords: female stress incontinence; Transobturator tension free vaginal tape TVTO
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid sling (Active Comparator): 70 patients with stress urinary incontinence treated with surgeon tailored hybrid sling
  Interventions: Procedure: Hybrid sling
- TVT-O (Active Comparator): 70 patients with stress urinary incontinence treated with conventional TVT-O
  Interventions: Procedure: TVT-O

INTERVENTIONS:
Procedure: Hybrid sling — sling formed of surgeon tailored autologous rectus sheath and polypropylene arms
  Arms: Hybrid sling
Procedure: TVT-O — midurethral transobturator vaginal tape
  Arms: TVT-O

SUMMARY:
a hybrid sling formed of a central part of autologus rectus sheath (2×6 cm) and two arms of polypropylene mesh (2×10cm) versus transobturator tension free vaginal tape(TVT-O)

DETAILED DESCRIPTION:
a surgeon tailored hybrid sling formed of a central part of autologus rectus sheath (2×6 cm) and two arms of polypropylene mesh (2×10cm) is used for treatment of urinary stree incontinence and its efficacy is compared to transobturator tension free vaginal tape (TVT-O) conventional mid urethral sling

ELIGIBILITY:
Inclusion Criteria:

* stress urinary incontinence

Exclusion Criteria:

* previous surgery for stress incontinence

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
cure rate | 1 year follow up
  negative cough stress test

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided